CLINICAL TRIAL: NCT04300140
Title: A Phase 1b/2 Study Of AVB-S6-500 In Combination With Cabozantinib, AVB-S6-500 In Combination With Cabozantinib and Nivolumab, and AVB-S6-500 Monotherapy in Patients With Advanced or Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Safety and Efficacy Study of AVB-S6-500 (Batiraxcept) in Patients With Advanced or Metastatic Clear Cell Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to business reasons
Sponsor: Aravive, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVB500-RCC-003
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Clear cell renal cell carcinoma; Renal cell carcinoma; Recurrent renal cell carcinoma; Kidney cancer; Kidney Neoplasms; Kidney Diseases; Urologic Neoplasms
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Kidney Diseases; Urologic Neoplasms | interventions — cabozantinib; VMBP protocol; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b: Batiraxcept + cabozantinib (Experimental): Two dose levels of batiraxcept administered Q2W (once every two weeks) in combination with QD (once a day) cabozantinib will be evaluated.
  Interventions: Drug: Batiraxcept; Drug: Cabozantinib (Cabo)
- Phase 2 Part A: batiraxcept + cabozantinib (Experimental): One dose level of batiraxcept administered Q2W in combination with QD cabozantinib will be evaluated.
  Interventions: Drug: Batiraxcept; Drug: Cabozantinib (Cabo)
- Phase 2 Part B: batiraxcept + cabozantinib + nivolumab (Experimental): One dose level of batiraxcept administered Q2W in combination with QD cabozantinib and nivolumab.
  Interventions: Drug: Batiraxcept; Drug: Cabozantinib (Cabo); Drug: Nivolumab
- Phase 2 Part C: batiraxcept alone (Experimental): One dose level of batiraxcept administered Q2W will be evaluated.
  Interventions: Drug: Batiraxcept

INTERVENTIONS:
Drug: Batiraxcept — Batiraxcept is experimental drug
  Other Names: AVB-S6-500
Drug: Cabozantinib (Cabo) — Cabozantinib is standard of care as monotherapy and in combination with nivolumab in ccRCC
  Other Names: Cabometyx®
  Arms: Phase 1b: Batiraxcept + cabozantinib; Phase 2 Part A: batiraxcept + cabozantinib; Phase 2 Part B: batiraxcept + cabozantinib + nivolumab
Drug: Nivolumab — Nivolumab is standard of care in the first line treatment of ccRCC
  Other Names: Opdivo®
  Arms: Phase 2 Part B: batiraxcept + cabozantinib + nivolumab

SUMMARY:
This is a Phase 1b/2 study of AVB-S6-500 designed to evaluate the safety and efficacy of AVB-S6-500 in combination with cabozantinib, AVB-S6-500 in combination with cabozantinib and nivolumab and AVB-S6-500 monotherapy in subjects with advanced or metastatic clear cell renal cell carcinoma (ccRCC). The phase 1b portion of the study is open label and patients with advanced ccRCC who had progressed on or after at least one prior line of treatment will receive AVB-S6-500 + cabozantinib. Two dose levels will be evaluated. The Phase 2 portion of the study is open-label 3-part study to evaluate efficacy and tolerability of AVB-S6-500 + cabozantinib, AVB-S6-500 + cabozantinib + nivolumab, and AVB-S6-500 alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologically confirmed advanced or metastatic clear cell Renal Cell Carcinoma confirmed by imaging. Phase 1b and Phase 2 Part A: has progressed on/after at least one front-line of treatment; Phase 2 Part B: No prior systemic treatment; Phase 2 Part C: not amenable to curative intent therapy.
* Must have radiologic imaging with a computed tomography (CT) scan or magnetic resonance imaging (MRI) within 28 days of enrollment
* Must have at least one measurable lesion according to RECIST 1.1
* ECOG performance status of 0-1
* Adequate bone marrow, liver and kidney function
* Life expectancy of >12 weeks
* At least 28 days between termination of prior major surgery or anticancer therapy or 14 days from last radiation therapy and administration of AVB-S6-500

Exclusion Criteria:

* Received prior treatment with cabozantinib (Phase1b and Phase 2 Part A)
* Received prior treatment with nivolumab (Phase 2 Part B)
* Concurrent anti-cancer therapy or any other interventional treatment or other interventional research trial
* History of prior malignancy within the past 3 years except adequately treated basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix or breast
* Symptomatic CNS metastasis or metastases
* Active GI disease that would impact absorption of cabozantinib
* Nephrotic range proteinuria at screening
* Evidence of pleural effusion, ascites etc that requires therapeutic intervention within 28 days prior to AVB-S6-500 administration
* Phase 2 Part A and Part B: Has had a major bleed in the last 3 months, uncontrolled hypertension despite treatment with antihypertensives or is not appropriate for treatment with cabozantinib in the Investigator's opinion
* Serious active infection requiring IV antibiotics and/or hospitalization at study entry
* Phase 2 Part B: Has active, known or suspected autoimmune disease, defined as requiring systemic treatment
* Active COVID-19, HIV, Hepatitis B or Hepatitis C virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events in Phase 1b as graded by NCI-CTCAE version 5.0 | 10 months
  Safety and tolerability of AVB-S6-500 in combination with cabozantinib.
Identify the recommended Phase 2 dose of AVB-S6-500 in combination with cabozantinib | 10 months
  Measured by dose limiting toxicities experienced in Phase 1b
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib (ORR) | 30 months
  Measured by objective response rate (ORR) in patients receiving AVB-S6-500 + cabozantinib in Phase 1b and Phase 2 Part A. ORR is proportion of subjects who have a partial or complete confirmed response to therapy relative to baseline as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib and nivolumab (ORR) | 30 months
  Measured by objective response rate (ORR) in patients receiving AVB-S6-500 + cabozantinib + nivolumab in Phase 2 Part B. ORR is proportion of subjects who have a partial or complete confirmed response to therapy relative to baseline as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Anti-tumor activity of AVB-S6-500 alone (ORR) | 30 months
  Measured by objective response rate (ORR) in patients receiving AVB-S6-500 in Phase 2 Part C. ORR is proportion of subjects who have a partial or complete confirmed response to therapy relative to baseline as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Anti-tumor activity of AVB-S6-500 alone (DOR) | 30 months
  Measured by duration of response (DOR) in patients receiving AVB-S6-500 in Phase 2 Part C. DOR is measured from the date of partial or complete response to therapy until the cancer progresses.
Anti-tumor activity of AVB-S6-500 alone (CBR) | 30 months
  Measured by clinical benefit rate (CBR) in patients receiving AVB-S6-500 in Phase 2 Part C. CBR is the proportion of subjects who have a complete or partial response to therapy or maintain stable disease.
Anti-tumor activity of AVB-S6-500 alone (PFS) | 30 months
  Measured by progression-free survival (PFS) in patients receiving AVB-S6-500 in Phase 2 Part C. PFS is the time from treatment until radiological disease progression or death.
Anti-tumor activity of AVB-S6-500 alone (OS) | 60 months
  Measured by overall survival (OS) in patients receiving AVB-S6-500 in Phase 2 Part C. OS is the time from the start of the treatment until death.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | 30 months
  Area under the AVB-S6-500 concentration-time curve.
Pharmacokinetics: Cmax | 30 months
  Maximum observed AVB-S6-500 concentration.
Pharmacokinetics: Tmax | 30 months
  Time of maximum observed AVB-S6-500 concentration.
Pharmacokinetics: t1/2 | 30 months
  Apparent terminal half-life of AVB-S6-500.
Pharmacodynamic marker assessment | 30 months
  Change from the baseline in GAS6 serum levels.
Anti-drug antibody (ADA) titers | 30 months
  Change from baseline in ADA titer.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib (CBR) | 30 months
  Measured by clinical benefit rate (CBR) in patients receiving AVB-S6-500 + cabozantinib in Phase 1b and Phase 2 Part A. CBR is the proportion of subjects who have a complete or partial response to therapy or maintain stable disease.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib (DOR) | 30 months
  Measured by duration of response (DOR) in patients receiving AVB-S6-500 in Phase 1b and Phase 2 Part A. DOR is measured from the date of partial or complete response to therapy until the cancer progresses.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib (OS) | 60 months
  Measured by overall survival (OS) in patients receiving AVB-S6-500 in Phase 1b and Phase 2 Part A. OS is the time from the start of the treatment until death.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib (PFS) | 30 months
  Measured by progression-free survival (PFS) in patients receiving AVB-S6-500 in Phase 1b and Phase 2 Part A, PFS is the time from treatment until radiological disease progression or death.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib and nivolumab (DOR) | 30 months
  Measured by duration of response (DOR) in patients receiving AVB-S6-500, cabozantinib and nivolumab in Phase 2 Part B. DOR is measured from the date of partial or complete response to therapy until the cancer progresses.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib and nivolumab (CBR) | 30 months
  Measured by clinical benefit rate (CBR) in patients receiving AVB-S6-500, cabozantinib and nivolumab in Phase 2 Part B. CBR is the proportion of subjects who have a complete or partial response to therapy or maintain stable disease.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib and nivolumab (PFS) | 30 months
  Measured by progression-free survival (PFS) in patients receiving AVB-S6-500, cabozantinib and nivolumab in Phase 2 Part B. PFS is the time from treatment until radiological disease progression or death.
Anti-tumor activity of AVB-S6-500 in combination with cabozantinib and nivolumab (OS) | 60 months
  Measured by overall survival (OS) in patients receiving AVB-S6-500, cabozantinib and nivolumab in Phase 2 Part B. OS is the time from the start of the treatment until death.
Incidence of adverse events in Phase 2 Part C as graded by NCI-CTCAE version 5.0 | 30 months
  Safety and tolerability of AVB-S6-500 alone
Incidence of adverse events in Phase 2 Part B as graded by NCI-CTCAE version 5.0 | 30 months
  Safety and tolerability of AVB-S6-500 in combination with cabozantinib and nivolumab

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Care of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Hollings Cancer Center (HCC), Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center (VICC), Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beckermann KE, Shah NJ, Campbell MT, Haas NB, Nelson A, Ornstein MC, Mao S, Keshava-Prasad HS, Hammers H, Gao X, Gourdin T, George S, Hoimes CJ, Hussain A, Jonasch E, Rini BI, Voss MH. Phase 1b/2 study of batiraxcept alone and in combination with cabozantinib with or without nivolumab for advanced clear cell renal cell carcinoma. Oncologist. 2025 Jun 4;30(6):oyaf138. doi: 10.1093/oncolo/oyaf138. PMID 40549043